CLINICAL TRIAL: NCT02822443
Title: The Impact of Integrating Emotion Focused Components Into Psychological Therapy
Brief Title: Improve: Integrating Emotion Focused Components Into Psychological Therapy
Acronym: Improve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNF100019_159425 /1
Record Dates: First submitted 2016-06-22; First posted 2016-07-04 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Unipolar Depression; Anxiety Disorder; Adjustment Disorder
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Adjustment Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAU - EFT (Experimental): This arm integrates emotion focused components (EFT; Greenberg, 2010) into psychological therapy (PT) as treatment-as-usual (TAU), aiming at clarifying and transforming maladaptive emotions. 25 (+/- 3) weekly sessions and up to three booster sessions of face-to-face outpatient psychotherapy; psychological therapy with focus on emotion-focused interventions.
  Interventions: Behavioral: Psychological therapy (PT) as TAU with integrated emotion focused components (TAU - EFT)
- TAU - SR (Experimental): This arm focuses on the training of self-regulation strategies (SR; Carver & Scheier, 2000) in the context of psychological therapy (PT) as treatment-as-usual (TAU). 25 (+/- 3) weekly sessions and up to three booster sessions of face-to-face outpatient psychotherapy; psychological therapy with focus on self-regulation without emotion-focused interventions.
  Interventions: Behavioral: Psychological therapy (PT) as TAU with focus on self-regulation (TAU - SR)

INTERVENTIONS:
Behavioral: Psychological therapy (PT) as TAU with integrated emotion focused components (TAU - EFT) — 25 (+/- 3) weekly sessions and up to three booster sessions of face-to-face outpatient psychotherapy; psychological therapy with focus on emotion-focused interventions.
  Arms: TAU - EFT
Behavioral: Psychological therapy (PT) as TAU with focus on self-regulation (TAU - SR) — 25 (+/- 3) weekly sessions and up to three booster sessions of face-to-face outpatient psychotherapy; psychological therapy with focus on self-regulation without emotion-focused interventions
  Arms: TAU - SR

SUMMARY:
The primary purpose of this study is to compare the efficacy of two treatment-as-usual (TAU) conditions: TAU with integration of emotion focused components (EFT) and TAU with focus on self-regulation (SR). Especially the long-term efficacy is evaluated with a focus on differential effects. Moreover, the mechanisms of change of both conditions are investigated.

DETAILED DESCRIPTION:
Background:

"General Psychotherapy" postulates an ongoing process of including all interventions and concepts relevant for a domain, be they from other approaches to psychotherapy or concepts from basic science. "Psychological Therapy" (PT) is a therapeutic approach largely corresponding to the ideas of General Psychotherapy. It draws mainly on empirically validated interventions from Cognitive Behavior Therapy (CBT) and is based on concepts with a strong basis in academic psychology and neighboring fields. PT is based on explicit individual case conceptualization, reference to general therapeutic factors, and an explicit prescriptive concept for building and maintaining the therapeutic relationship. However the range of emotion-related interventions commonly used in PT is limited when compared with an approach like Emotion Focused Therapy (EFT). EFT appears thus as a suitable complement and enrichment to PT as commonly practiced. However, effects of integrating EFT-based interventions in a way that is close to common integrative practice have not yet been studied.

Objective:

To compare the efficacy of two treatment-as-usual (TAU) conditions: TAU with integration of EFT components and TAU with focus on self-regulation (SR).

Methods:

In Switzerland, a randomized-controlled trail will be carried out in secondary care, comparing the efficacy of TAU - EFT and TAU - SR for adults with major depressive disorder, anxiety disorder or adjustment disorder. Respondents will be followed until 36 months after end of therapy (measures will be taken at baseline, after 8 and after 16 weeks, at the end of therapy after 25 weeks, 6 months, 12 months and 36 months follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder, Anxiety Disorder or Adjustment Disorder according to DSM-IV as main diagnosis
* Minimum age of 18 years
* Mastery of the German language for being able to undergo a psychotherapy in German
* Written informed consent to participate voluntary in the study

Exclusion Criteria:

* Acute suicidality or immediate threats of self-harm
* Diagnosis or history of a psychotic disorder
* Mood incongruent psychotic symptoms
* Bipolar disorder
* Comorbid chronic organic disorder
* Substance use disorder as a main diagnosis
* Indication for a residential treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptom impairment measured by the Brief Symptom Inventory (BSI; Franke, 2000) | After 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Change from baseline in depressive symptoms measured by the Beck Depression Inventory (BDI-II; Hautzinger et al., 2006) | After 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Change from baseline in anxiety symptoms measured by the Beck Anxiety Inventory (BAI; Ehlers & Margraf, 2007) | After 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up

SECONDARY OUTCOMES:
Severity of panic disorder and agoraphobia with the Panic and Agoraphobia Scale (PAS; Bandelow, 1997) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Severity of social phobia measured by the Social Phobia Scale SPS; Stangier et al., 1999) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Severity of social interaction anxiety measured by the Social Interaction Anxiety Scale (SIAS; Stangier et al., 1999) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Severity of anxiety symptoms measured by the Questionnaire for General Anxiety Disorder (GAD-7; Spitzer et al., 2006) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Psychological well-being measured with the WHO Well-Being Index (WHO-5; Henkel et al., 2004) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Health-related quality of life measured with the Short Form Healthy Survey (SF-12; Gandek et al., 1998) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Motivational schemata measured by the Questionnaire for Analysis of Motivational Schemata (FAMOS; grosse Holtforth & Grawe, 2000) | Baseline, end of therapy after 25 weeks
Motivational incongruence measured by the Incongruence Questionnaire (K-INK; grosse Holtforth et al., 2003) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Interpersonal problems measured by the Inventory of Interpersonal Problems (IIP-32; Thomas et al., 2011) | Baseline, after 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Personality structure measured by the Operationalized Psychodynamic Diagnosis Structure Questionnaire (OPD-SFK; Ehrenthal et al., 2012) | Baseline, end of therapy after 25 weeks
Personality traits measured by the Inventory of Personality Organization (IPO-16; Zimmermann et al., 2013) | Baseline
Ambivalence over emotional expressiveness measured by the Ambivalence over the Expression of Emotion Scale (AVEX; Trachsel et al., 2010) | Baseline, end of therapy after 25 weeks
Emotional competency measured by the Questionnaire for the self-assessment of emotional competencies (SEK-27; Berking & Znoj, 2008) | Baseline, end of therapy after 25 weeks
Generalized expectancies for negative mood regulation measured by the Negative Mood Regulation Scale (NMR-SF; Pfeiffer et al., 2013) | Baseline, end of therapy after 25 weeks
Psychological flexibility measured by the Acceptance and Action Questionnaire (Fragebogen zu Akzeptanz und Handeln; FAH-II; Gloster et al., 2013) | Baseline, end of therapy after 25 weeks
General self-efficacy measured by the General Self-Efficacy Scale (SWE; Schwarzer & Jerusalem, 1999) | Baseline, end of therapy after 25 weeks
Therapy evaluation and outcome expectancies measured by the Patient Questionnaire on Therapy Expectation and Evaluation (PATHEV; Schulte, 2005) | Baseline
Social desirability measured by the Balanced Inventory of Desirable Responding (BIDR-K; Winkler et al., 2006) | Baseline
Client satisfaction measured by the Brief Global Measure of Client Satisfaction (ZUF-8; Schmidt & Wittmann, 2002) | After 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
External assessment of interpersonal personality measured by the Impact Message Inventory (IMI-R; Caspar et al. 2002) | Baseline, end of therapy after 25 weeks
External assessment of resources measured by the Bernese Inventory of Resources (REF-F and REF-T; Tröske, 2000) | Baseline, end of therapy after 25 weeks
External assessment of positive interpersonal qualities measured by the Inventory of Interpersonal Strengths (IIS; Hatcher & Rogers, 2012) | Baseline, end of therapy after 25 weeks
Goal attainment measured by the Goal Attainment Scaling (GAS; Kirusek, 1994) | After 8 weeks, after 16 weeks, end of therapy after 25 weeks, 6 months follow-up, 12 months follow-up and 36 months follow-up
Regular quality monitoring with the Bern Post Session Report, Patient and Therapist Version (BPSR-P/T; Flückiger et al. 2010) | Weekly until 25 weeks
Symptom impairment measured by the Symptom Checklist (SCL-9; Bogerts et al., 2001) | Weekly until 25 weeks
Implicit motives measured by the Picture-Story-Exercise - Online Version (PSE-O: Bernecker & Jobst, 2013) | Baseline, end of therapy after 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franz Caspar, Prof. PhD, Principal Investigator — University of Bern, Switzerland
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babl A, Grosse Holtforth M, Heer S, Lin M, Stahli A, Holstein D, Belz M, Egenolf Y, Frischknecht E, Ramseyer F, Regli D, Schmied E, Fluckiger C, Brodbeck J, Berger T, Caspar F. Psychotherapy integration under scrutiny: investigating the impact of integrating emotion-focused components into a CBT-based approach: a study protocol of a randomized controlled trial. BMC Psychiatry. 2016 Nov 24;16(1):423. doi: 10.1186/s12888-016-1136-7. PMID 27881113